CLINICAL TRIAL: NCT00857324
Title: A Phase I/II, Multi-Center, Open Label Study of Vorinostat Plus Melphalan and Prednisone (ZMP) in Advanced, Refractory Multiple Myeloma Patients
Brief Title: Study of Vorinostat Plus Melphalan and Prednisone (Zmp) in Advanced, Refractory Multiple Myeloma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Phase I of the study was completed, but Phase 2 has not been activated
Sponsor: Tiziana Marangon (Other)
Responsible Party: Sponsor-Investigator, Tiziana Marangon, Sponsor, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZMP-1; 2008-000646-32
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
Keywords: Refractory or relapsed patients; dose-finding; Vorinostat
MeSH Terms: conditions — Multiple Myeloma | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZMP (Experimental): Combination with Vorinostat, Melphalan and Prednisone
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Patients will start induction treatment with a standard dose of MP and escalating doses of Vorinostat:
  * Melphalan 0.18 mg/Kg for 4 days; Prednisone 1.5 mg/Kg for 4 days. Each cycle will be repeated every 28 days for a total of 6 courses
  * In the first part of the study, the standard oral MP will be combined with escalating doses of Vorinostat.
  Level -1 Vorinostat = 100 mg daily on days 1-21 Melphalan = 0.18 mg/kg on days 1 - 4 Prednisone = 1.5 mg/kg on days 1 - 4
  Level 0 Vorinostat = 200 mg daily on days 1-21 Melphalan = 0.18 mg/kg on days 1 - 4 Prednisone = 1.5 mg/kg on days 1 - 4
  Level +1 Vorinostat = 300 mg daily on days 1-21 Melphalan = 0.18 mg/kg on days 1 - 4 Prednisone = 1.5 mg/kg on days 1 - 4
  Level +2 Vorinostat = 400 mg daily on days 1-21 Melphalan = 0.18 mg/kg on days 1 - 4 Prednisone = 1.5 mg/kg on days 1 - 4

SUMMARY:
The purpose of this study is to determine whether the association of ZMP is safe and provides benefits in patients with relapsed/refractory MM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal for 24 consecutive months or surgically sterilized or agree to continuous abstinence from heterosexual sexual contact or willing to use effective contraception for 4 weeks prior to beginning study drug therapy, during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of therapy; female patients not pregnant or nursing; female with a negative pregnancy test.
* Male patient agrees to use an acceptable method for contraception during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of Vorinostat therapy.
* Patient was previously diagnosed with symptomatic MM based on standard criteria, and has measurable disease.
* Patient is relapsed or refractory after a minimum of 3 weeks from prior therapies (patients must have recovered from toxicities related to prior therapies).
* Patient has a Karnofsky performance status ≥ 60%.
* Patient has a life-expectancy > 3 months.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness or social situation that would prevent the subject from signing the informed consent form or limit the compliance with study medications and requirements.
* Pregnant or beast feeding females.
* Use of any other concomitant standard/experimental anti-myeloma drug or therapy.
* Known positive for HIV or active infectious hepatitis, type B or C.
* Known congenital long QT syndrome.
* Ongoing therapy with anti-arrhythmic drugs or other medicinal products which led to QT prolongation and cumulative high dose of anthracycline.
* Any clinically significant illness that would, in the investigator's opinion, increase the patient's risk for toxicity. Patients has not plasmacell leukaemia defined as the presence of more than 20% plasma cells in the peripheral blood and an absolute plasma cell count of at least 2000/uL.
* Patients has not a currently active malignancy, except non melanoma skin cancer and carcinoma in situ of the cervix. Patients should not be considered to have a currently active second malignancy if they have completed therapy for a prior malignancy and are disease free from prior malignancies for >5 years and are considered by their physicians to be at less then 30% risk of relapse
* History of allergic reactions related to study drugs.
* Prior exposure to HDACi. Patients exposed to valproic acid could be eligible with a wash out period of at least 30 days.
* Patients scheduled to undergo autologous or allogenic bone marrow transplant within 4 week of the initiation of Vorinostat administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The dose limiting toxicity (DLT)of Vorinostat with MP | one year
The maximum tolerated dose (MTD) of Vorinostat in association with MP | 1 year
A significant number of PR or higher (>40%) following the proposed ZMP therapy | 1 year

SECONDARY OUTCOMES:
Duration of Progression Free Survival | 5 Years
Duration of Overall Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Principal Investigator — University of Turin, Italy
Locations (4):
- Italy (4):
  - Dipartimento Medicina Clinica e Sperimentale, Padua
  - A.O.U. S. Giovanni Battista, Torino
  - Policlinico Universitario di Udine, Udine
  - Azienda Ospedaliera di Verona - Policlinico G.B. Rossi, Verona